CLINICAL TRIAL: NCT00389350
Title: The Effect of an Extract of Green Tea on Glucose Control in Adults With Type 2 Diabetes
Brief Title: Effect of an Extract of Green Tea on Adults With Type 2 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Todd MacKenzie, Principle Investigator, Professor, Data Science, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hitchcock Tea 1
Record Dates: First submitted 2006-10-16; First posted 2006-10-18 (Estimated); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Tea

INTERVENTIONS:
Drug: Extract of Green and Black Tea
  Other Names: Placebo Arm

SUMMARY:
The objective of this study was to determine if taking an extract of green tea for three months could improve glucose control in adults with diabetes.

DETAILED DESCRIPTION:
Background: Recent evidence suggests that tea from Camellia Senensis (e.g., green, oolong and black tea) may have a hypoglycemic effect.

Objective: We evaluated the ability of an extract of green and black tea to improve glucose control over a three month period using a double blinded randomized multiple dose (either placebo, 375mg or 750mg) study in adults in with Type 2 Diabetes.

Patients: The 49 subjects who completed this study were predominantly whites with an average age of 65, a median duration of Diabetes of 6 years, and 80% reported using hypoglycemic medication.

Measurements: HbA1c at three months was the primary endpoint. Results: After three months the mean changes in HbA1c were +0.4, +0.3 and +0.5, in the placebo, 375mg and 750mg arms, respectively. The changes were not significantly different between study arms.

Limitations: Evaluation of a particular extract that contained components of black teas as well as green tea. Power insufficient to detect changes in HbA1c < 0.5.

Conclusions: We did not find a hypoglycemic effect of extract of green tea in adults with Type 2 Diabetes, but cannot rule out the possibility that tea may have a small beneficial effect.

ELIGIBILITY:
Inclusion Criteria:

* Adults with Diabetes not taking insulin

Exclusion Criteria:

* pregnancy, warfarin therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2005-08; Study Completion 2006-06

PRIMARY OUTCOMES:
HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Todd A MacKenzie, PhD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States